CLINICAL TRIAL: NCT01835925
Title: Rectal Cancer Consortium: BrUOG 285: A Comprehensive Program to Identify Therapeutic Targets and Develop Targeted Agents for Testing With Total Neoadjuvant Treatment for Stage II-III Rectal Cancer BrUOG= Brown University Oncology Research Group
Brief Title: Rectal Cancer Consortium
Status: Completed | Type: Observational
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Other Study IDs: 285
Record Dates: First submitted 2013-04-09; First posted 2013-04-19 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Rectal Cancer
Keywords: adenocarcinoma of rectum; rectal cancer; stage II; stage III
MeSH Terms: conditions — Rectal Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimen from diagnosis from rectal cancer
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tissue specmien
  Interventions: Genetic: Tissue specimen

INTERVENTIONS:
Genetic: Tissue specimen

SUMMARY:
The purpose of this study is to study which genes are abnormal in rectal cancer and see if this predicts how well chemotherapy and radiation will reduce the size of cancer and whether cancer recurs after surgery.

DETAILED DESCRIPTION:
Specific gene mutations have become targets for specific therapies. For example lung adenocarcinomas with an EGFR (epidermal growth factor receptor) mutation can be targeted with an EGFR tyrosine kinase inhibitor achieve striking and durable responses and improved survival. Another example is the identification of the echinoderm microtubule-associated protein-like 4/anaplastic lymphoma kinase (ALK) gene fusions which have led to significant therapeutic gains in the small percentage of patients with lung adenocarcinoma whose cancers exhibit this mutation. Specific mutations have been found in colon cancer and specific drugs targeting these gene alterations are in development. As future therapeutic protocols specific for these mutations are developed, patients who agree may be notified of their eligibility for these studies.

The aims of this study are to link mutational analyses with clinical outcome. It is recommended that patients receive 8 cycles of mFOLFOX6 (modified FOLFOX) and 50.4 Gy radiation with concurrent fluoropyrimidine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven adenocarcinoma of the rectum with no evidence of distant metastases.
* The tumor must be clinically Stage II (T3-4 N0) or III (T1-4 N1-2).
* Patients must have no evidence of distant metastases including liver metastases, peritoneal seeding, or inguinal lymphadenopathy.
* Patients who completed or are actively enrolled in the CONTRE study and patients undergoing treatment for rectal cancer following the TNT (Total Neoadjuvant Treatment) format (see below) for whom sufficient tissue is available for the required research analyses may be enrolled in this study retroactively.
* For those who have not yet received treatment for rectal adenocarcinoma, these patients must not have received prior chemotherapy or pelvic radiation for rectal cancer, or prior pelvic radiation for any other malignancy that would prevent the patient from receiving the required radiation treatments for this study.
* Patients must not have an active concurrent invasive malignancy other than non-melanoma skin cancers. Patients with malignancies diagnosed within 5 years prior to randomization which have been effectively treated and are deemed to be at low risk for recurrence are eligible.
* Patients must be > 18 years of age, ECOG (performance status) 0-1.
* ANC (absolute neutrophil count) >1,500/µl, platelets >100,000/µl, total bilirubin <2.0 mg/dl or direct bilirubin <1.0 mg/dl, alkaline phosphatase <3xULN, ALT <3xULN, creatinine <1.5xULN.
* Signed informed consent; able to comply with study and/or follow- up procedures
* Peripheral neuropathy < grade 1.
* The intention of the treating physicians is to administer Total Neoadjuvant Treatment as per the suggested treatment guidelines in section 4 and section 5 or as per standard institutional policies.

Exclusion Criteria:

* Evidence of metastatic disease.
* Rectal cancers other than adenocarcinoma, i.e., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, cloacogenic carcinoma, etc.
* Pregnancy or lactation at the time of proposed randomization. Eligible patients of reproductive potential (both sexes) must agree to use adequate contraception.
* Synchronous invasive colon cancer.
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the patient from receiving any chemotherapy treatment option or would prevent required follow-up.
* Patients with active inflammatory bowel disease, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0 or other serious medical illness which might limit the ability of the patient to receive protocol therapy.
* Known hypersensitivity to 5-fluorouracil or oxaliplatin
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Insufficient tumor tissue available for the required genomic analyses and patient unable or unwilling to undergo repeat examination and biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II or III rectal cancer (adenocarcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Tumor tissue to predict likelihood of achieving pathologic complete response post standard treatment. | baseline

SECONDARY OUTCOMES:
Tumor tissue results with clinical outcome post standard treatment. . | annually for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island